CLINICAL TRIAL: NCT04910893
Title: Cytokine Adsorption in Severe, Refractory Septic Shock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: CytoSorbents Europe GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Cytosorb
Record Dates: First submitted 2021-05-27; First posted 2021-06-02 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Septic Shock; Cytokine Storm
Keywords: Septic Shock; Cytokine Adsorption; Hemadsorption; extracorporeal removal
MeSH Terms: conditions — Shock, Septic; Cytokine Release Syndrome | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Prospective interventional study with comparative matched septic shock cohort
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cytokine Adsorption Arm (Experimental): Intervention with CytoSorb
  Interventions: Device: Cytokine Adsorption
- Historical Comparison (Other): Patients extracted from a septic shock population treated at the same institution between 2010 and 2018 and matched to the intervention group.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: Cytokine Adsorption — Cytokine adsorption therapy will be provided continuously for 72 hours by means of the CytoSorb® (CytoSorbents Corporation, Monmouth Junction, USA) column, run in series to a veno-venous continuous hemodialysis system, which will be exchanged every 24 hours.
  Other Names: CytoSorb
  Arms: Cytokine Adsorption Arm
Other: Standard of Care — Standard intensive care of patients suffering septic shock
  Arms: Historical Comparison

SUMMARY:
Septic shock and the underlying dysregulated inflammatory host-response remain a major contributor to mortality in critically ill patients. Cytokine adsorption represents an attractive approach to the treatment of septic shock. Nevertheless, its effect on circulating cytokine levels, as well as on the course of disease remains largely unassessed.

DETAILED DESCRIPTION:
Cytokine-release plays an important role in the physiology of immune response to pathologic influences by recruiting immune cells to the pathogenic loci, be they of infectious or of non-infectious nature. Once at the focus, the activated immune cells can in turn release more cytokines if a more extensive immune response is needed. This extremely important mechanism for the organism, can however become pathological if the positive feedback loop between immune cells and cytokines, for any reason, overshoots in form of a so called cytokine storm and substantial amounts of released cytokines gain a systemic influence. The acute complication of this immune over-reaction is a SIRS, which can critically escalate into a potentially lethal multiple organ dysfunction syndrome, thus requiring immediate intensive care treatment.

It is, having this framework in mind, the reason why the CytoSorb-Adsorber has been developed as a new therapeutic milestone. Essentially a haemoperfusion-filter, which through its layering with polymer beads (Divinylbenzene/ Polyvinylpyrrolidone) can adsorb cytokines as well as multiple inflammatory mediators and thus effectively remove them from the bloodstream, reducing their possible systemic influence and hence improving the outcome for patients being treated with it.

The CytoSorb-Adsorber is an already CE-approved product, which has demonstrated its capacity to significantly reduce cytokine-levels such as IL-6, IL-8, IL-10, TNFα, HMGB-1, IL-1ra in a variety of pre-clinical studies. As well as in a clinical randomised multicentre study, which tested the CytoSorb-Adsorber on a cohort of ALI/ ARDS and severely septic/ septically shocked patients. The results of the later study can be very positively assessed, first of all and most importantly showing, that no security concerns had to be had in regard to the haemoperfusion-filter, as no adverse-effects attributable to the device were found. And further, by proving an effect on systemic cytokine-levels in form of a significant reduction in IL-6, IL-8, MCP-1 and IL-1ra, as well as a reduction in mortality of those patients with high initial cytokine levels, effectively reducing the 60 day mortality rate from 60% to 17% in a pool of 14 patients.

With the intention to further elucidate the usefulness and clinical importance of this device this study proposes a prospective recruitment of patients in severe refractory septic shock to test the efficiency of this device.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed septic shock in the 24 hours ensuing diagnosis:

(I) severe, refractory septic shock defined as:

1. an acute SOFA score increase ≥2 points consequent to a presumed or proven infection
2. volume resuscitation of at least 30ml/kg in the last 24 hours
3. a Vasopressor Dependency Index11 (VPI) above or equal to 3
4. a persistently elevated serum lactate level >2mmol/l (II) Interleukin-6 levels equal or above 1000 ng/l (III) were above 18 years of age.

Exclusion Criteria:

1. Contraindication on ethical grounds
2. child bearing or breastfeeding women
3. terminal patients
4. human immunodeficiency virus with a CD4 cell count <0.2 106/l
5. allergy to Polystyrene/ Divinylbenzene, Polycarbonate, Polypropylene, Silicon or Polyester
6. need for extra-corporeal membrane oxygenation
7. no given consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-11-27 (Actual); Primary Completion 2018-08-24 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in circulating Interleukin-6 levels over time | Mixed Model Assessment at timepoints 0, 24, 48, 72 hours
  Change in circulating Interleukin-6 levels, stratified by groups, over the initial 72 hours ensuing fulfillment of inclusion criteria
Change in Vasopressor requirements over time | Mixed Model Assessment at timepoints 0, 2, 4, 8, 12 , 24, 48, 72 hours
  Change in the Vasopressor Dependency Index, stratified by groups, over the initial 72 hours ensuing fulfillment of inclusion criteria
Cumulative intensive care mortality at 30 days | 30 days post fulfillment of inclusion criteria
  Intensive care mortality assessment at day 30 between groups

SECONDARY OUTCOMES:
Change in C-reactive protein levels over time | Mixed Model Assessment at timepoints 0, 24, 48, 72 hours
  Change in C-reactive protein levels, stratified by groups, over the initial 72 hours ensuing fulfillment of inclusion criteria
Change in Procalcitonin levels over time | Mixed Model Assessment at timepoints 0, 24, 48, 72 hours
  Change in Procalcitonin levels, stratified by groups, over the initial 72 hours ensuing fulfillment of inclusion criteria
Change in SOFA Score over time | Mixed Model Assessment at timepoints 0, 24, 48, 72 hours
  Change in SOFA Score, stratified by groups, over the initial 72 hours ensuing fulfillment of inclusion criteria
Change in arterial lactate levels over time | Mixed Model Assessment at timepoints 0, 2, 4, 8, 12 , 24, 48, 72 hours
  Change in arterial lactate levels, stratified by groups, over the initial 72 hours ensuing fulfillment of inclusion criteria
Change in cardiac index over time | Mixed Model Assessment at timepoints 0, 2, 4, 8, 12 , 24, 48, 72 hours
  Change in cardiac index, stratified by groups, over the initial 72 hours ensuing fulfillment of inclusion criteria
Change in Extra Vascular Lung Water Index over time | Mixed Model Assessment at timepoints 0, 24, 48, 72 hours
  Change in Extra Vascular Lung Water Index, stratified by groups, over the initial 72 hours ensuing fulfillment of inclusion criteria
Change in daily Infused Volume over time | Mixed Model Assessment at timepoints 0, 24, 48, 72 hours
  Change in daily Infused Volume, stratified by groups, over the initial 72 hours ensuing fulfillment of inclusion criteria
Change in PaO2/ FiO2 Ratio over time | Mixed Model Assessment at timepoints 0, 2, 4, 8, 12 , 24, 48, 72 hours
  Change in PaO2/ FiO2 Ratio, stratified by groups, over the initial 72 hours ensuing fulfillment of inclusion criteria
Change in Serum Albumin levels over time | Mixed Model Assessment at timepoints 0, 24, 48, 72 hours
  Change in Serum Albumin levels, stratified by groups, over the initial 72 hours ensuing fulfillment of inclusion criteria
Change in Bilirubin levels over time | Mixed Model Assessment at timepoints 0, 24, 48, 72 hours
  Change in Bilirubin levels, stratified by groups, over the initial 72 hours ensuing fulfillment of inclusion criteria

CONTACTS AND LOCATIONS:
Overall Officials: Marco Maggiorini, MD, Principal Investigator — Medizinische Intensivstation D-HOER 27, UniversitatsSpital Zürich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang H, Ma S. The cytokine storm and factors determining the sequence and severity of organ dysfunction in multiple organ dysfunction syndrome. Am J Emerg Med. 2008 Jul;26(6):711-5. doi: 10.1016/j.ajem.2007.10.031. PMID 18606328
- [Background] Taniguchi T. Cytokine adsorbing columns. Contrib Nephrol. 2010;166:134-141. doi: 10.1159/000314863. Epub 2010 May 7. PMID 20473001
- [Background] Morris C, Gray L, Giovannelli M. Early report: The use of Cytosorb haemabsorption column as an adjunct in managing severe sepsis: initial experiences, review and recommendations. J Intensive Care Soc. 2015 Aug;16(3):257-264. doi: 10.1177/1751143715574855. Epub 2015 Mar 18. PMID 28979423
- [Background] Rimmele T, Kellum JA. Clinical review: blood purification for sepsis. Crit Care. 2011;15(1):205. doi: 10.1186/cc9411. Epub 2011 Feb 16. PMID 21371356
- [Background] Reiter K, Bordoni V, Dall'Olio G, Ricatti MG, Soli M, Ruperti S, Soffiati G, Galloni E, D'Intini V, Bellomo R, Ronco C. In vitro removal of therapeutic drugs with a novel adsorbent system. Blood Purif. 2002;20(4):380-8. doi: 10.1159/000063108. PMID 12169849
- [Background] Kellum JA, Song M, Venkataraman R. Hemoadsorption removes tumor necrosis factor, interleukin-6, and interleukin-10, reduces nuclear factor-kappaB DNA binding, and improves short-term survival in lethal endotoxemia. Crit Care Med. 2004 Mar;32(3):801-5. doi: 10.1097/01.ccm.0000114997.39857.69. PMID 15090965
- [Background] Peng ZY, Carter MJ, Kellum JA. Effects of hemoadsorption on cytokine removal and short-term survival in septic rats. Crit Care Med. 2008 May;36(5):1573-7. doi: 10.1097/CCM.0b013e318170b9a7. PMID 18434884
- [Background] D Schädler, C Porzelius, A Jörres, G Marx, A Meier-Hellmann, C Putensen, M Quintel, C Spies, C Engel, NWeiler, M Kuhlmann. A multicenter randomized controlled study of an extracorporeal cytokine hemoadsorption device in septic patients. Critical Care 2013, 17(Suppl 2):P62 (19 March 2013).